CLINICAL TRIAL: NCT01441635
Title: Phase 2a Proof Of Concept Study to Evaluate the Safety and Efficacy of Elagolix in Pre-Menopausal Women With Heavy Uterine Bleeding and Uterine Fibroids
Brief Title: Safety and Efficacy of Elagolix in Pre-Menopausal Women With Heavy Uterine Bleeding and Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-663
Record Dates: First submitted 2011-09-06; First posted 2011-09-28 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Heavy Uterine Bleeding; Uterine Fibroids
Keywords: Uterine Fibroids; Heavy Uterine Bleeding; Elagolix; Menorrhagia; ABT-620; Leiomyomata; Elagolix sodium
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — elagolix; Estradiol; Norethindrone Acetate; estradiol, norethindrone drug combination; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort 4 Elagolix 400 mg QD (Experimental): Participants received elagolix 400 mg once a day (QD) for 3 months.
  Interventions: Drug: Elagolix
- Cohort 4 Elagolix 100 mg BID (Experimental): Participants received elagolix 100 mg twice a day (BID) for 3 months.
  Interventions: Drug: Elagolix
- Cohort 4 Placebo (Placebo Comparator): Participants received placebo to elagolix BID for 3 months.
  Interventions: Drug: Placebo
- Cohort 1 Elagolix 200 mg BID (Experimental): Participants received elagolix 200 mg twice a day for 3 months.
  Interventions: Drug: Elagolix
- Cohort 1 Placebo (Placebo Comparator): Participants received placebo to elagolix twice a day for 3 months.
  Interventions: Drug: Placebo
- Cohort 3 Elagolix 200 mg BID + LD E2/NETA (Placebo Comparator): Participants received elagolix 200 mg twice a day plus continuous low-dose (LD) estradiol (E2) 0.5 mg/norethindrone acetate 0.1 mg (NETA) once a day for 3 months.
  Interventions: Drug: Elagolix; Drug: Estradiol/Norethindrone acetate (E2/NETA)
- Cohort 5 Elagolix 600 mg QD (Experimental): Participants received elagolix 600 mg once a day for 3 months.
  Interventions: Drug: Elagolix
- Cohort 2 Elagolix 300 mg BID (Experimental): Participants received elagolix 300 mg twice a day for 3 months.
  Interventions: Drug: Elagolix
- Cohort 2 Placebo (Experimental): Participants received placebo to elagolix BID for 3 months.
  Interventions: Drug: Placebo
- Cohort 6 Elagolix 300 mg BID + CEP (Experimental): Participants received elagolix 300 mg twice a day plus cyclical estrogen/progesterone (CEP, consisting of estradiol 1 mg a day and progesterone 200 mg on days 17 to 28 of each 30-day treatment cycle) for 3 months.
  Interventions: Drug: Elagolix; Drug: Estradiol; Drug: Progesterone

INTERVENTIONS:
Drug: Elagolix — Elagolix tablets
  Other Names: ABT-620
  Arms: Cohort 1 Elagolix 200 mg BID; Cohort 2 Elagolix 300 mg BID; Cohort 3 Elagolix 200 mg BID + LD E2/NETA; Cohort 4 Elagolix 100 mg BID; Cohort 4 Elagolix 400 mg QD; Cohort 5 Elagolix 600 mg QD; Cohort 6 Elagolix 300 mg BID + CEP
Drug: Placebo — Matching placebo tablets
  Arms: Cohort 1 Placebo; Cohort 2 Placebo; Cohort 4 Placebo
Drug: Estradiol/Norethindrone acetate (E2/NETA) — A continuous once-daily oral tablet containing estrogen and progestin; the low-dose strength contains estradiol 0.5 mg and norethindrone acetate 0.1 mg.
  Other Names: Activella®
  Arms: Cohort 3 Elagolix 200 mg BID + LD E2/NETA
Drug: Estradiol — 1.0 mg micronized estradiol tablets administered once a day
  Other Names: Estrace®
  Arms: Cohort 6 Elagolix 300 mg BID + CEP
Drug: Progesterone — Progesterone 200 mg administered during the last 12 days of the 28-day menstrual cycle
  Other Names: Prometrium®
  Arms: Cohort 6 Elagolix 300 mg BID + CEP

SUMMARY:
The purpose of this proof-of-concept study is to assess the safety and effectiveness of elagolix versus placebo to reduce uterine bleeding associated with uterine fibroids, and to reduce fibroid volume and uterine volume in premenopausal women 20 to 49 years of age with heavy uterine bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a pre-menopausal female 20 to 49 years of age.
* Subject has a diagnosis of uterine fibroids documented by a pelvic ultrasound assessed by a central reader and verification that a fibroid present met the following criteria:

  * At least 1 fibroid with diameter ≥ 2 cm (longest diameter), or multiple small fibroids with a total uterine volume of ≥ 200 cm³ to ≤ 2,500 cm³ (approximately 22 weeks' gestation) as documented by a centrally read ultrasound.
  * Only intramural, submucosal non-pedunculated, and subserosal fibroids qualified subjects for enrollment (intracavitary pedunculated fibroids were exclusionary).
  * Ultrasound procedures were performed during the Screening Period, and subjects were not randomized until the investigator reviewed the central reader results verifying the inclusion requirements.
* Subject has a history of regular menstrual cycles between 24 to 35 days.
* Subject has heavy uterine bleeding associated with uterine fibroids as evidenced by blood loss > 80 mL during 2 screening menstrual cycles, measured by the alkaline hematin method.

Exclusion Criteria:

* Subject has had a myomectomy, uterine artery embolization, or high intensity focused ultrasound for fibroid destruction within 1 year prior to randomization or any history of endometrial ablation.
* Subject has a history of osteoporosis or other metabolic bone disease.
* Subject shows evidence of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric (including depression), or neurologic diseases or any uncontrolled medical illness such as uncontrolled type 2 diabetes.
* Subject has a history of clinically significant condition(s) including but not limited to:

  * Endometriosis
  * Epilepsy or seizures
  * Type 1 diabetes
  * Any cancer (except basal cell carcinoma of the skin), including breast or ovarian cancer or subject has taken any systemic cancer chemotherapy

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2011-09-08 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Archer DF, Stewart EA, Jain RI, Feldman RA, Lukes AS, North JD, Soliman AM, Gao J, Ng JW, Chwalisz K. Elagolix for the management of heavy menstrual bleeding associated with uterine fibroids: results from a phase 2a proof-of-concept study. Fertil Steril. 2017 Jul;108(1):152-160.e4. doi: 10.1016/j.fertnstert.2017.05.006. Epub 2017 Jun 1. PMID 28579415
- [Derived] Coyne KS, Soliman AM, Margolis MK, Thompson CL, Chwalisz K. Validation of the 4 week recall version of the Uterine Fibroid Symptom and Health-related Quality of Life (UFS-QOL) Questionnaire. Curr Med Res Opin. 2017 Feb;33(2):193-200. doi: 10.1080/03007995.2016.1248382. Epub 2016 Nov 18. PMID 27733082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 271 female participants were enrolled into the study across 45 sites in the United States.
Pre-assignment Details: Six cohorts of participants were enrolled, with 3 double-blind cohorts comparing elagolix with placebo, 2 open-label cohorts assessing add-back therapies, and 1 open-label cohort assessing the elagolix 600 mg QD dosing regimen.
Period: Overall Study
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Started | 32 | 33 | 16 | 35 | 18 | 34 | 30 | 30 | 16 | 27
Completed | 26 | 27 | 13 | 28 | 16 | 29 | 24 | 26 | 14 | 25
Not Completed | 6 | 6 | 3 | 7 | 2 | 5 | 6 | 4 | 2 | 2
Not completed — Adverse Event | 4 | 3 | 1 | 5 | 1 | 2 | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 1
Not completed — Noncompliance | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Surgery or Invasive Intervention | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Received Exclusionary Medication | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP | Total
Number analyzed (Participants) | 32 | 33 | 16 | 35 | 18 | 34 | 30 | 30 | 16 | 27 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (5.50) | 42.1 (5.09) | 41.1 (5.88) | 43.1 (4.29) | 44.0 (4.24) | 40.9 (6.02) | 40.8 (5.78) | 42.6 (5.55) | 41.6 (7.10) | 41.6 (5.26) | 41.8 (5.4)
Age, Customized [Count of Participants; unit: Participants]
  < 35 years | 7 | 3 | 2 | 2 | 0 | 5 | 4 | 3 | 3 | 3 | 32
  35 to < 40 years | 6 | 5 | 5 | 5 | 2 | 8 | 6 | 5 | 3 | 6 | 51
  40 to < 45 years | 8 | 13 | 2 | 13 | 7 | 10 | 11 | 9 | 3 | 10 | 86
  ≥ 45 years | 11 | 12 | 7 | 15 | 9 | 11 | 9 | 13 | 7 | 8 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 16 | 35 | 18 | 34 | 30 | 30 | 16 | 27 | 271
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 8 | 1 | 1 | 1 | 1 | 6 | 0 | 2 | 12 | 33
  Not Hispanic or Latino | 31 | 25 | 15 | 34 | 17 | 33 | 24 | 30 | 14 | 15 | 238
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 10 | 3 | 7 | 3 | 7 | 5 | 6 | 6 | 11 | 63
  Black | 25 | 23 | 13 | 28 | 14 | 26 | 24 | 23 | 9 | 15 | 200
  Asian | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Multirace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to the Last 28 Days of Treatment in Menstrual Blood Loss (MBL)
Description: The alkaline hematin method was used for the assessment of MBL. Sanitary products were collected at screening and for any spotting or bleeding episodes that occurred during treatment.
  Participants with missing MBL volume for the last treatment period and no bleeding indicated in the electronic daily bleeding diary (eDiary) in the last treatment period, and participants with no post-baseline MBL data were assigned an MBL value of zero.
Time Frame: Baseline (last menstrual cycle during the screening period) and the last 28 days of treatment (approximately days 61 to 90)
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants, excluding participants with less than 28 days of treatment. Last observation carried forward (LOCF) imputation was used for participants with no MBL volume reported by alkaline hematin method but with light to heavy bleeding reported in the eDiary.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 31 | 31 | 15 | 32 | 18 | 33 | 28 | 30 | 15 | 26
mL
  Baseline | 213.70 (108.08) | 269.36 (163.17) | 321.73 (327.57) | 335.11 (322.68) | 251.72 (160.29) | 247.70 (177.72) | 215.62 (122.84) | 206.27 (125.08) | 349.17 (424.12) | 257.99 (207.33)
  Change from Baseline | -183.97 (132.19) | -184.69 (187.05) | -10.46 (85.04) | -272.97 (271.39) | -79.00 (161.33) | -192.33 (191.51) | -189.05 (151.15) | -202.57 (127.93) | -175.31 (342.14) | -216.15 (157.08)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -205.9, 95% CI 2-sided [-295.77 to -116.01], Standard Error of Mean 45.10
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -189.9, 95% CI 2-sided [-278.33 to -101.53], Standard Error of Mean 44.36
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -138.0, 95% CI 2-sided [-220.18 to -55.76], Standard Error of Mean 40.86
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p = 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -130.6, 95% CI 2-sided [-206.70 to -54.60], Standard Error of Mean 37.68

2. Secondary Outcome: Percent Change From Baseline to the Last 28 Days of Treatment in Menstrual Blood Loss (MBL)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants, excluding participants with less than 28 days of treatment. Last observation carried forward (LOCF) imputation was used for participants with no MBL volume reported by alkaline hematin method but with light to heavy bleeding reported in the electronic diary.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 31 | 31 | 15 | 32 | 18 | 33 | 28 | 30 | 15 | 26
percent change | -83.83 (35.23) | -71.85 (49.20) | -6.98 (40.78) | -81.03 (55.77) | -11.12 (103.11) | -79.60 (43.63) | -88.58 (39.58) | -97.31 (12.57) | -42.64 (39.68) | -85.39 (28.08)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -75.60, 95% CI 2-sided [-102.93 to -48.28], Standard Error of Mean 13.71
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -64.27, 95% CI 2-sided [-91.14 to -37.39], Standard Error of Mean 13.48
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.005, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -67.67, 95% CI 2-sided [-113.39 to -21.96], Standard Error of Mean 22.73
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS mean Difference = -56.84, 95% CI 2-sided [-73.24 to -40.45], Standard Error of Mean 8.12

3. Secondary Outcome: Percentage of Participants With MBL < 80 mL and With a ≥ 50% Reduction From Baseline in MBL During the Last 28 Days of Treatment
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants, excluding participants with less than 28 days of treatment. LOCF imputation was used for participants with no MBL volume reported by alkaline hematin method but with light to heavy bleeding reported in the eDiary.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 31 | 31 | 15 | 33 | 18 | 33 | 28 | 30 | 15 | 26
percentage of participants | 84 | 74 | 13 | 85 | 17 | 85 | 93 | 97 | 33 | 85
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p < 0.001, Fisher Exact

4. Secondary Outcome: Percentage of Participants With MBL < 80 mL During the Last 28 Days of Treatment
Description: as for outcome 1
Time Frame: The last 28 days of treatment (approximately days 61 to 90)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 31 | 31 | 15 | 33 | 18 | 33 | 28 | 30 | 15 | 26
percentage of participants | 84 | 74 | 13 | 85 | 22 | 88 | 93 | 97 | 47 | 88
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Elagolix 100 mg BID; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p < 0.001, Fisher Exact

5. Secondary Outcome: Percentage of Participants With a ≥ 50% Reduction From Baseline in MBL During the Last 28 Days of Treatment
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 31 | 31 | 15 | 33 | 18 | 33 | 28 | 30 | 15 | 26
percentage of participants | 84 | 74 | 13 | 91 | 28 | 85 | 93 | 97 | 40 | 88
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p < 0.001, Fisher Exact

6. Secondary Outcome: Percentage of Participants With No Change, Decrease From Baseline, or Increase From Baseline in Hemoglobin at Month 3
Description: The percentage of subjects with changes in hemoglobin concentration from Baseline to Month 3 in each of the following categories:
  * No change from baseline in hemoglobin
  * Decrease from baseline in hemoglobin ≥ -0.5 g/dL
  * Decrease from baseline in hemoglobin ≥ -1.0 g/dL
  * Increase from baseline in hemoglobin ≥ 0.5 g/dL
  * Increase from baseline in hemoglobin ≥ 1.0 g/dL
  The above categories are not all mutually exclusive or exhaustive.
Time Frame: Baseline and Month 3
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available hemoglobin data.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 23 | 24 | 11 | 27 | 14 | 28 | 23 | 25 | 14 | 21
percentage of participants
  No Change | 0 | 0 | 9 | 0 | 0 | 0 | 4 | 0 | 0 | 5
  Decreases from -0.5 to 0 g/dL | 9 | 17 | 0 | 4 | 21 | 14 | 4 | 0 | 21 | 5
  Decreases from -1.0 to -0.5 g/dL | 4 | 4 | 27 | 11 | 14 | 0 | 4 | 0 | 7 | 10
  Increase ≥ 0.5 g/dL | 78 | 71 | 18 | 67 | 29 | 75 | 83 | 76 | 29 | 71
  Increase ≥ 1.0 g/dL | 61 | 71 | 9 | 59 | 29 | 43 | 57 | 52 | 29 | 62

7. Secondary Outcome: Change in Hemoglobin Concentration From Baseline to Month 3
Time Frame: Baseline and Month 3
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available hemoglobin data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 23 | 24 | 11 | 27 | 14 | 28 | 23 | 25 | 14 | 21
g/dL | 1.18 (0.99) | 1.30 (1.19) | -0.43 (1.28) | 1.13 (1.29) | 0.28 (1.33) | 0.92 (0.81) | 1.40 (1.18) | 1.19 (0.85) | 0.31 (1.20) | 1.54 (1.81)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = 1.8, 95% CI 2-sided [0.97 to 2.56], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = 1.8, 95% CI 2-sided [1.00 to 2.56], Standard Error of Mean 0.39
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.024, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = 0.9, 95% CI 2-sided [0.13 to 1.75], Standard Error of Mean 0.40
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p = 0.005, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = 0.9, 95% CI 2-sided [0.28 to 1.51], Standard Error of Mean 0.30

8. Secondary Outcome: Change From Baseline to Month 3 in Uterine Bleeding Score
Description: Participants recorded the previous days' presence and severity of bleeding every morning in an electronic diary (eDiary) according to the Mansfield-Voda-Jorgenson Menstrual Bleeding Scale:
  * 1 (Spotting): A drop or 2 of blood, not even requiring sanitary protection.
  * 2 (Very light): Needing to change the least absorbent tampon or pad 1 to 2 times per day.
  * 3 (Light): Needing to change a low or regular absorbency tampon or pad 2 or 3 times per day.
  * 4 (Moderate): Needing to change a regular absorbency tampon or pad every 3 to 4 hours.
  * 5 (Heavy): Needing to change a high absorbency tampon or pad every 3 to 4 hours.
  * 6 (Very heavy/gushing): Very heavy bleeding, protection hardly works at all; needing to change the highest absorbency tampon or pad every hour or 2.
Time Frame: Baseline (average bleeding score over the 30 days prior to first dose) and month 3 (average bleeding score over days 61 to 90)
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available bleeding score data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 30 | 30 | 15 | 32 | 17 | 32 | 26 | 27 | 15 | 25
units on a scale | -0.50 (0.56) | -0.37 (0.46) | -0.19 (0.33) | -0.52 (0.65) | -0.22 (0.32) | -0.24 (0.47) | -0.44 (0.71) | -0.53 (0.33) | -0.38 (0.77) | -0.25 (0.64)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p = 0.011, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -0.36, 95% CI 2-sided [-0.63 to -0.08], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p = 0.030, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -0.31, 95% CI 2-sided [-0.59 to -0.03], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.109, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -0.26, 95% CI 2-sided [-0.59 to 0.06], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p = 0.002, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -0.50, 95% CI 2-sided [-0.80 to -0.19], Standard Error of Mean 0.15

9. Secondary Outcome: Change From Baseline to Month 3 in Percentage of Days With Any Uterine Bleeding
Description: Participants recorded the previous days' presence and severity of bleeding every morning in an electronic diary (eDiary) according to the Mansfield-Voda-Jorgenson Menstrual Bleeding Scale:
  * 1 (Spotting): A drop or 2 of blood, not even requiring sanitary protection.
  * 2 (Very light): Needing to change the least absorbent tampon or pad 1 to 2 times per day.
  * 3 (Light): Needing to change a low or regular absorbency tampon or pad 2 or 3 times per day.
  * 4 (Moderate): Needing to change a regular absorbency tampon or pad every 3 to 4 hours.
  * 5 (Heavy): Needing to change a high absorbency tampon or pad every 3 to 4 hours.
  * 6 (Very heavy/gushing): Very heavy bleeding, protection hardly works at all; needing to change the highest absorbency tampon or pad every hour or 2.
  A day with any uterine bleeding is defined as a days with a bleeding score ≥ 1.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 30 | 30 | 15 | 32 | 17 | 32 | 26 | 27 | 15 | 25
percentage of days | -15.22 (14.77) | -11.00 (15.52) | -5.78 (10.58) | -15.82 (17.88) | -6.99 (12.82) | 3.63 (24.74) | -15.38 (23.21) | -16.91 (11.13) | -13.95 (23.83) | 1.73 (26.09)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Elagolix 100 mg BID; Test type: Superiority; p = 0.020, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -10.29, 95% CI 2-sided [-18.90 to -1.67], Standard Error of Mean 4.32
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p = 0.087, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -7.62, 95% CI 2-sided [-16.36 to 1.13], Standard Error of Mean 4.39
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.045, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -8.81, 95% CI 2-sided [-17.43 to -0.19], Standard Error of Mean 4.28
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p = 0.002, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -13.69, 95% CI 2-sided [-22.06 to -5.32], Standard Error of Mean 4.14

10. Secondary Outcome: Change From Baseline to Month 3 in Percentage of Days With Moderate to Very Heavy Bleeding
Description: Participants recorded the previous days' presence and severity of bleeding every morning in an electronic diary (eDiary) according to the Mansfield-Voda-Jorgenson Menstrual Bleeding Scale:
  * 1 (Spotting): A drop or 2 of blood, not even requiring sanitary protection.
  * 2 (Very light): Needing to change the least absorbent tampon or pad 1 to 2 times per day.
  * 3 (Light): Needing to change a low or regular absorbency tampon or pad 2 or 3 times per day.
  * 4 (Moderate): Needing to change a regular absorbency tampon or pad every 3 to 4 hours.
  * 5 (Heavy): Needing to change a high absorbency tampon or pad every 3 to 4 hours.
  * 6 (Very heavy/gushing): Very heavy bleeding, protection hardly works at all; needing to change the highest absorbency tampon or pad every hour or 2.
  A day with moderate to very heavy bleeding is defined as a days with a bleeding score ≥ 3.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 30 | 30 | 15 | 32 | 17 | 32 | 26 | 27 | 15 | 25
percentage of days | -7.22 (9.27) | -5.00 (7.87) | -4.00 (5.37) | -7.03 (10.89) | -3.08 (5.88) | -7.92 (6.43) | -6.15 (8.47) | -8.02 (5.41) | -3.31 (10.40) | -6.80 (10.69)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Placebo; Test type: Superiority; p = 0.008, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -5.51, 95% CI 2-sided [-9.56 to -1.47], Standard Error of Mean 2.03
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p = 0.020, ANCOVA; LS Mean Difference = -4.95, 95% CI 2-sided [-9.11 to -0.80], Standard Error of Mean 2.08
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.194, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -3.63, 95% CI 2-sided [-9.18 to 1.91], Standard Error of Mean 2.75
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p = 0.001, ANCOVA; ANCOVA model with treatment as a factor and baseline as a covariate; LS Mean Difference = -7.20, 95% CI 2-sided [-11.33 to -3.07], Standard Error of Mean 2.04

11. Secondary Outcome: Percentage of Participants With Any Uterine Bleeding or Moderate to Very Heavy Uterine Bleeding at Month 3
Description: Participants recorded the previous days' presence and severity of bleeding every morning in an eDiary according to the Mansfield-Voda-Jorgenson Menstrual Bleeding Scale:
  * 1 (Spotting): A drop or 2 of blood, not even requiring sanitary protection.
  * 2 (Very light): Needing to change the least absorbent tampon or pad 1 to 2 times per day.
  * 3 (Light): Needing to change a low or regular absorbency tampon or pad 2 or 3 times per day.
  * 4 (Moderate): Needing to change a regular absorbency tampon or pad every 3 to 4 hours.
  * 5 (Heavy): Needing to change a high absorbency tampon or pad every 3 to 4 hours.
  * 6 (Very heavy/gushing): Very heavy bleeding, protection hardly works at all; needing to change the highest absorbency tampon or pad every hour or 2.
  Any bleeding is defined as a score ≥ 1 and moderate to very heavy bleeding is defined as a score ≥ 3.
Time Frame: Month 3 (average bleeding score over days 61 to 90)
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available bleeding score data at month 3.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 30 | 30 | 15 | 32 | 17 | 32 | 26 | 27 | 15 | 26
percentage of participants
  Any bleeding | 37 | 57 | 93 | 47 | 94 | 78 | 27 | 26 | 80 | 69
  Moderate to Very Heavy Bleeding | 27 | 40 | 87 | 28 | 82 | 31 | 15 | 7 | 73 | 35

12. Secondary Outcome: Percentage of Participants With Suppression of Bleeding (Spotting Allowed) or Amenorrhea During the Last 56 Days of Treatment
Description: Suppression of bleeding is defined as no record of bleeding (spotting allowed) in the e-diary and no record of bleeding Indicated in the alkaline hematin data during the last 56 days of treatment.
  Amenorrhea is defined as no record of bleeding or spotting indicated in the e-diary and no record of bleeding or spotting Indicated in the alkaline hematin data during the last 56 days of treatment.
Time Frame: The last 56 days of treatment (approximately days 33 to 90)
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants including participants with less than 56 days of treatment who bled but excluded those who did not bleed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 30 | 29 | 15 | 32 | 18 | 32 | 26 | 29 | 16 | 26
percentage of participants
  Suppression of bleeding | 66 | 45 | 0 | 66 | 0 | 31 | 77 | 79 | 0 | 32
  Amenorrhea | 60 | 31 | 0 | 44 | 0 | 19 | 73 | 66 | 0 | 19

13. Secondary Outcome: Percent Change From Baseline to Month 3 in Uterine Volume
Description: Uterine volume was determined using transabdominal ultrasound. The images were analyzed by a central imaging center.
Time Frame: Baseline and month 3
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available uterine volume data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 22 | 20 | 9 | 22 | 12 | 22 | 20 | 20 | 12 | 11
percent change | -21.01 (26.79) | -21.37 (24.84) | 18.72 (15.59) | -21.68 (29.80) | -8.62 (20.58) | -17.43 (19.51) | -27.99 (23.34) | -33.25 (16.55) | -1.92 (17.52) | -10.06 (30.93)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Elagolix 100 mg BID; Test type: Superiority; p < 0.001, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p < 0.001, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.052, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p < 0.001, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor

14. Secondary Outcome: Percentage of Participants With ≥ 25% Reduction in Uterine Volume at Month 3 / Final Visit
Description: Uterine volume was determined using transabdominal ultrasound. The images were analyzed by a central imaging center.
Time Frame: Baseline and month 3 or the final visit during the treatment period for participants who prematurely discontinued.
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 30 | 30 | 15 | 31 | 18 | 33 | 27 | 29 | 15 | 24
percentage of participants | 53 | 43 | 7 | 48 | 11 | 42 | 56 | 69 | 7 | 25
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Elagolix 100 mg BID; Test type: Superiority; p = 0.003, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p = 0.016, Fisher Exact
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.012, Fisher Exact
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p < 0.001, Fisher Exact

15. Secondary Outcome: Percent Change From Baseline to Month 3 in Volume of the Largest Fibroid
Description: The volume of the largest fibroid was determined using transabdominal ultrasound. The images were analyzed by a central imaging center.
Time Frame: Baseline and month 3
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available fibroid volume data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 19 | 18 | 9 | 22 | 12 | 22 | 18 | 20 | 12 | 10
percent change | 14.23 (187.83) | -22.19 (51.14) | -7.26 (36.35) | -38.52 (41.72) | -2.05 (71.83) | -25.77 (46.64) | -16.60 (39.61) | -35.79 (24.49) | 6.70 (45.42) | -4.94 (100.68)
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Elagolix 100 mg BID; Test type: Superiority; p = 0.161, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p = 0.173, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.072, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p = 0.003, Kruskal-Wallis; One-way Kruskal-Wallis test with treatment as a factor

16. Secondary Outcome: Percentage of Participants With ≥ 25% Reduction in Volume of Largest Fibroid at Month 3 / Final Visit
Description: as for outcome 15
Time Frame: Baseline and month 3 or the final visit during the treatment period for participants who prematurely discontinued.
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 28 | 29 | 15 | 31 | 17 | 33 | 25 | 29 | 15 | 21
percentage of participants | 57 | 52 | 33 | 68 | 35 | 58 | 60 | 55 | 27 | 48
Statistical Analysis 1: Comparison: Cohort 4 Elagolix 400 mg QD vs Cohort 4 Elagolix 100 mg BID; Test type: Superiority; p = 0.203, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 4 Elagolix 100 mg BID vs Cohort 4 Placebo; Test type: Superiority; p = 0.342, Fisher Exact
Statistical Analysis 3: Comparison: Cohort 1 Elagolix 200 mg BID vs Cohort 1 Placebo; Test type: Superiority; p = 0.038, Fisher Exact
Statistical Analysis 4: Comparison: Cohort 2 Elagolix 300 mg BID vs Cohort 2 Placebo; Test type: Superiority; p = 0.111, Fisher Exact

17. Secondary Outcome: Change From Baseline to Month 3 in the Uterine Fibroid Symptom Quality of Life Questionnaire (UFS-QoL)
Description: The UFS-QoL is a disease-specific, self-administered, validated questionnaire developed to evaluate the symptoms associated with uterine fibroids and their impact on health-related quality of life (HRQL) in women with symptomatic uterine fibroids. The questionnaire consists of 37 questions, divided into 2 parts: 1) an 8-item symptom severity scale and 2) a 29-item HRQL subscale comprising 6 domains (concern, activities, energy/mood, control, self-consiousness, and sexual function), with a 4-week recall. All items are scored on a 5-point scale, ranging from "not at all" to "a very great deal" for symptom severity items and "none of the time" to "all of the time" for the HRQL items. Symptom severity and HRQL subscale scores were summed and transformed into a 0 to 100 point scale to provide a total score for each of the 2 components.
  Lower symptom severity scores indicate better quality of life and higher total HRQL scores indicate better quality of life.
Time Frame: Baseline and month 3
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available UFS-QoL data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 23 | 21 | 9 | 26 | 13 | 22 | 20 | 25 | 13 | 14
units on a scale
  Symptom severity | -39.0 (24.70) | -33.2 (28.17) | -19.6 (32.80) | -31.6 (28.87) | -21.4 (20.63) | -20.3 (25.35) | -36.4 (24.74) | -44.1 (22.12) | -12.0 (22.49) | -39.1 (24.09)
  HRQL total: number analyzed (Participants) | 22 | 21 | 9 | 25 | 13 | 22 | 20 | 25 | 13 | 14
  HRQL total | 35.3 (21.87) | 29.1 (30.96) | 16.3 (30.43) | 36.0 (27.91) | 18.3 (36.66) | 28.6 (24.12) | 29.9 (30.72) | 33.5 (29.42) | 11.0 (20.90) | 33.1 (30.34)

18. Secondary Outcome: Change From Baseline to Month 3 in the Uterine Fibroids Daily Symptom Scale Scores
Description: The uterine fibroid daily symptom scale is self-administered questionnaire, with a scale that ranges from 0 to 10 for the symptoms of pelvic pain, fatigue, and cramping and the impact of uterine fibroids on the subject's daily life, with 0 being the absence of the symptom and 10 being the worst severity of the symptoms or completely preventing the subjects from performing daily activities. Participants self-reported values daily in the e-Diary.
Time Frame: Baseline (average score over the 30 days prior to first dose) and month 3 (average score over days 61 to 90)
Population: Randomized (Cohorts 1, 2, and 4) or treated (Cohorts 3, 5, and 6) participants with available data at baseline and month 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 18 | 18 | 9 | 18 | 11 | 22 | 16 | 20 | 9 | 11
units on a scale
  Pelvic pain | -1.0 (2.27) | -0.2 (2.39) | -0.3 (1.45) | -0.6 (1.75) | -1.4 (1.62) | -1.1 (1.35) | -0.9 (2.15) | -1.0 (1.75) | -1.2 (1.73) | -2.4 (3.00)
  Fatigue | -0.5 (1.26) | -0.0 (2.23) | -0.6 (1.45) | -0.6 (1.29) | -0.5 (1.69) | -1.2 (1.92) | -1.0 (2.57) | -1.5 (1.16) | -0.5 (2.88) | -2.1 (3.11)
  Menstrual cramping | -1.2 (1.31) | -0.7 (2.51) | -0.5 (1.55) | -0.9 (1.16) | -1.2 (0.80) | -0.9 (1.25) | -1.1 (1.35) | -1.2 (1.09) | -1.0 (2.33) | -1.3 (2.15)
  Impact of uterine fibroids | -1.1 (1.18) | -0.4 (1.86) | -0.8 (1.40) | -1.0 (1.37) | -1.0 (1.81) | -0.9 (1.62) | -1.7 (2.41) | -1.3 (1.11) | -1.0 (2.18) | -3.1 (2.78)

19. Secondary Outcome: Change From Baseline to Month 3 in the Subject Surgery Intention Questionnaire (SSIQ) Version 2.0
Description: The Subject Intention Questionnaire (SSIQ) is a non-validated, exploratory questionnaires intended to evaluate the subject's intent to undergo surgical procedures if current endometriosis-associated symptoms continued. The scoring scale ranged from 0 (not at all likely to consider surgery) to 10 (very likely to consider surgery).
  SSIQ included the 2 following questions:
  1. How likely are you to consider having myomectomy surgery to treat your uterine fibroid if your symptoms continue as they are now?
  2. How likely are you to consider hysterectomy surgery if your uterine fibroid symptoms continue as they are now?
Time Frame: Baseline and month 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 23 | 21 | 9 | 9 | 6 | 22 | 20 | 25 | 13 | 14
units on a scale
  Likelihood of having myomectomy | -1.2 (3.68) | -3.1 (4.52) | 1.0 (2.12) | -1.8 (4.70) | 2.3 (5.35) | -1.4 (4.34) | -1.7 (4.18) | -0.6 (5.10) | 0.4 (4.16) | 0.1 (2.63)
  Likelihood of having hysterectomy: number analyzed (Participants) | 23 | 20 | 9 | 9 | 6 | 22 | 20 | 25 | 13 | 14
  Likelihood of having hysterectomy | 0.0 (4.04) | -1.9 (4.19) | 2.0 (3.64) | -0.8 (4.91) | -0.3 (0.52) | -0.7 (3.10) | -0.8 (4.42) | 0.2 (3.65) | 0.0 (1.96) | -1.5 (3.92)

20. Secondary Outcome: Change From Baseline to Month 3 in the Physician Surgery Intention Questionnaire (PSIQ) Version 2.0
Description: The Physician Intention Questionnaire (PSIQ) is a non-validated, exploratory questionnaire intended to evaluate the investigator's intent to recommend surgical procedures if current endometriosis-associated symptoms continued. The scoring scale ranged from 0 (not at all likely to recommend surgery) to 10 (very likely to recommend surgery).
  The PSIQ included the 2 following questions:
  1. How likely are you to recommend myomectomy to treat this patient's uterine fibroid if her symptoms continue as they are now?
  2. How likely are you to recommend definitive surgery hysterectomy for this patient if her uterine fibroid symptoms continue as they are now?
Time Frame: Baseline and month 3
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 4 Elagolix 400 mg QD | Cohort 4 Elagolix 100 mg BID | Cohort 4 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 1 Placebo | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 5 Elagolix 600 mg QD | Cohort 2 Elagolix 300 mg BID | Cohort 2 Placebo | Cohort 6 Elagolix 300 mg BID + CEP
Number analyzed (Participants) | 23 | 21 | 9 | 9 | 7 | 22 | 20 | 24 | 13 | 14
units on a scale
  Likelihood to recommend myomectomy | -0.9 (2.86) | -1.3 (3.31) | -2.7 (3.53) | -0.8 (1.76) | 0.7 (1.11) | -0.6 (2.97) | -1.3 (3.62) | -1.2 (3.59) | 0.0 (3.25) | 0.0 (3.94)
  Likelihood to recommend hysterectomy | -0.8 (3.34) | -1.8 (4.37) | -0.2 (3.15) | -2.2 (2.82) | 0.4 (1.62) | -1.4 (3.08) | -2.3 (3.99) | -1.5 (3.96) | -0.6 (2.81) | -2.8 (2.98)

ADVERSE EVENTS:
Time Frame: From the date of the first dose of study drug through up to 30 days after the last dose of study drug, up to 4 months.
Groups:
- Cohort 4 Golix 400 mg QD: Participants received elagolix 400 mg once a day (QD) for 3 months.
Arm/Group | Cohort 1 Placebo | Cohort 1 Elagolix 200 mg BID | Cohort 2 Placebo | Cohort 2 Elagolix 300 mg BID | Cohort 3 Elagolix 200 mg BID + LD E2/NETA | Cohort 4 Placebo | Cohort 4 Elagolix 100 mg BID | Cohort 4 Golix 400 mg QD | Cohort 5 Elagolix 600 mg QD | Cohort 6 Elagolix 300 mg BID + CEP
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/35 | 0/16 | 0/30 | 0/34 | 0/16 | 0/33 | 0/32 | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/35 | 0/16 | 1/30 | 0/34 | 2/16 | 2/33 | 0/32 | 2/30 | 0/27
Other Adverse Events (participants affected / at risk) | 8/18 | 26/35 | 10/16 | 20/30 | 20/34 | 9/16 | 20/33 | 24/32 | 22/30 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Placebo (N=18) | Cohort 1 Elagolix 200 mg BID (N=35) | Cohort 2 Placebo (N=16) | Cohort 2 Elagolix 300 mg BID (N=30) | Cohort 3 Elagolix 200 mg BID + LD E2/NETA (N=34) | Cohort 4 Placebo (N=16) | Cohort 4 Elagolix 100 mg BID (N=33) | Cohort 4 Golix 400 mg QD (N=32) | Cohort 5 Elagolix 600 mg QD (N=30) | Cohort 6 Elagolix 300 mg BID + CEP (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0
NECROSIS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
ABORTION INDUCED (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Placebo (N=18) | Cohort 1 Elagolix 200 mg BID (N=35) | Cohort 2 Placebo (N=16) | Cohort 2 Elagolix 300 mg BID (N=30) | Cohort 3 Elagolix 200 mg BID + LD E2/NETA (N=34) | Cohort 4 Placebo (N=16) | Cohort 4 Elagolix 100 mg BID (N=33) | Cohort 4 Golix 400 mg QD (N=32) | Cohort 5 Elagolix 600 mg QD (N=30) | Cohort 6 Elagolix 300 mg BID + CEP (N=27)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 | 3 (5) | 0 | 0 | 0 | 0 | 2 (2) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 0 | 3 (4) | 2 (2) | 2 (2) | 0 | 1 (1) | 0 | 5 (5) | 9 (9) | 4 (4)
FATIGUE (General disorders) | 1 (1) | 2 (2) | 0 | 0 | 4 (4) | 0 | 1 (1) | 4 (4) | 2 (2) | 0
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
BRONCHITIS (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
VAGINITIS BACTERIAL (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2)
WEIGHT INCREASED (Investigations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 | 2 (3) | 0 | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 1 (1) | 0 | 3 (3) | 0 | 0 | 0 | 2 (2) | 0
DIZZINESS (Nervous system disorders) | 0 | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 0 | 1 (1) | 3 (3) | 6 (6) | 0
HEADACHE (Nervous system disorders) | 0 | 3 (3) | 3 (3) | 6 (6) | 5 (5) | 0 | 3 (3) | 4 (4) | 9 (11) | 2 (2)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MOOD SWINGS (Psychiatric disorders) | 1 (1) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 2 (2)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (2) | 2 (2) | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 3 (3) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 2 (3) | 0 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 1 (1) | 19 (20) | 3 (3) | 15 (15) | 9 (9) | 2 (2) | 15 (16) | 20 (21) | 15 (15) | 5 (5)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 2 (2) | 0 | 0 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (2) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 3 (3) | 3 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (2) | 0 | 0 | 0 | 0 | 2 (2) | 0
CHILLS (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
IRRITABILITY (General disorders) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
VESSEL PUNCTURE SITE PAIN (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
VULVOVAGINITIS (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
SPIDER VEIN (Vascular disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 (3) | 0 | 0 | 0 | 0 | 0
LIBIDO DECREASED (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
AMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
BREAST CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
FURUNCLE (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
INFECTED BITES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 2 (2) | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 3 (3) | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 1 (1) | 2 (3) | 0
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 2 (2) | 1 (1) | 0 | 0
DYSPAREUNIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 0 | 0
CHLOASMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 3 (3) | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.